CLINICAL TRIAL: NCT07081464
Title: Study of the Impact of Locus Coeruleus Dysfunction on Cognitive Function in Young Subjects With Ondine Syndrome
Brief Title: Locus Coeruleus and CCHS (Congenital Central Hypoventilation Syndrome)
Acronym: ONDINE-LC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241606; N° IDRCB : 2025-A00156-43 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ondine Syndrome (Congenital Central Hypoventilation Syndrome)
Keywords: Locus Coeruleus; PHOX2B; Cognitive Dysfunction; EEG; Pupillometry; MRI; Ondine Syndrome
MeSH Terms: conditions — Sleep Apnea, Central; Congenital central hypoventilation syndrome; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with severe Ondine syndrome (PHOX2B mutation with ≥ 27 alanine expansions)
  Interventions: Other: MRI, EEG, Pupillometry
- Subjects with moderate Ondine syndrome (PHOX2B mutation with < 27 alanine expansions);
  Interventions: Other: MRI, EEG, Pupillometry

INTERVENTIONS:
Other: MRI, EEG, Pupillometry — Comparison of P300 wave amplitude, pupillometric responses, functional and structural brain connectivity, socio-adaptive function, cardiac autonomic balance between two phenotypic severity groups of young patients with Ondine Syndrome.

SUMMARY:
This study investigates whether cognitive dysfunction in young patients with congenital central hypoventilation syndrome (Ondine Syndrome) is related to the severity of the disease and dysfunction of the locus coeruleus (a brainstem structure involved in autonomic control and cognition). The investigators will assess cognitive evoked potentials (P300 wave) using high-resolution EEG during attention tasks, pupillometry, brain MRI, neuropsychological tests, and heart rate variability. Patients with different severities of PHOX2B gene mutation (alanine expansions <27 vs. ≥27) will be compared.

DETAILED DESCRIPTION:
Ondine Syndrome (congenital central hypoventilation syndrome) is a rare autosomal dominant genetic disorder caused by mutations in PHOX2B. Patients require lifelong nocturnal ventilation and often have cognitive impairments. The cause of cognitive deficits is uncertain: possible hypoxic brain injury or direct effects of PHOX2B mutations on brain regions like the locus coeruleus.

This cross-sectional study includes 21 patients aged 7-20 years with Ondine Syndrome and PARM-type (polyalanine repeat mutation) PHOX2B mutations, divided into moderate (<27 alanine expansions) and severe (≥27 expansions) groups. During routine hospitalization, participants undergo:

High-resolution EEG with evoked potentials during auditory and visual attention tasks to measure P300 wave amplitude.

Pupillometry during the same tasks to assess locus coeruleus function.

3T (3 Tesla magnetic resonance imaging) MRI (anatomical and diffusion imaging) without sedation.

Neuropsychological assessment with the Vineland test.

Holter ECG to analyze heart rate variability.

The goal is to link locus coeruleus dysfunction to disease severity and explore its impact on cognition, autonomic balance, and sleep."

ELIGIBILITY:
Inclusion Criteria:

* Neonatal diagnosis of Ondine Syndrome.
* PARM-type PHOX2B mutation.
* Age 7 to 20 years.
* Receiving nocturnal ventilation.
* Consent obtained. Affiliated with social security.

Exclusion Criteria:

* Severe autism spectrum disorder preventing test completion.
* Legal guardianship or curatorship.

Ages: 7 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Minors and young adults aged 7 to 20 years diagnosed neonatally with Ondine Syndrome, carrying a PARM-type PHOX2B mutation and requiring nocturnal ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the P300 wave (peak-to-baseline) recorded by high-resolution EEG during visual and auditory attention tasks. | 24 hours
  Measurement of cognitive evoked potential P300 amplitude using a 64-electrode EEG system during Flanker and oddball paradigms to assess locus coeruleus function.

SECONDARY OUTCOMES:
Ratio of maximal pupil diameter during attention tasks to resting pupil diameter measured by pupillometry. | 24 hours
Functional connectivity parameters of the locus coeruleus measured by high-resolution EEG and 3T brain MRI diffusion imaging. | 24 hours
Scores of socio-adaptive behavior from the Vineland neuropsychological test (Vineland Adaptative Behavior Scales II, with scores ranging from 20 to 160; higher scores indicating better functioning). | 24 hours
  Vineland Adaptative Behavior Scales II, with scores ranging from 20 to 160; higher scores indicating better functioning.
Heart rate variability parameters from Holter ECG monitoring. | 24 hours
Structural connectivity parameters of the locus coeruleus measured by high-resolution EEG and 3T brain MRI diffusion imaging. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier MAUVAIS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, Ap-hp / DRCI, France